CLINICAL TRIAL: NCT03459560
Title: Effectiveness of Polypill for Primary Prevention of Cardiovascular Disease (PolyPars): Study Design and Rationale for a Pragmatic Cluster Randomized Controlled Trial
Brief Title: Prevention of Cardiovascular Disease With Polypill Among Pars Cohort Participants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MOH-700/107
Record Dates: First submitted 2018-03-03; First posted 2018-03-09 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Cardiovascular Diseases
Keywords: fixed-dose combination therapy; Polypill; Prevention; Cardiovascular diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PolyPill (Experimental): Single daily dose of PolyPill and minimal care.
  Interventions: Drug: PolyPill
- Control (No Intervention): Only minimal care

INTERVENTIONS:
Drug: PolyPill — After the baseline enrollment and excluding non-eligible participants, we randomized villages to Polypill and control arms. Follow-ups are scheduled for 1, 3, and 6 months after the initial enrollment in the Polypill arm and every six months thereafter. For the minimal care arm, the follow-ups are arranged every six months.
  Other Names: PolyPill-E, Polypill-V
  Arms: PolyPill

SUMMARY:
The purpose of this study is to determine the effects of a fixed dose combination of enalapril (or valsartan), with hydrochlorthiazide, atorvastatin and acetylsalicylic acid (PolyPill) on primary and secondary prevention of cardiovascular disease in participants of Pars Cohort of Iran.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVDs) are the most common causes of death and disability in Iran and account for nearly half of all-cause mortality in Iranians. Therefore, prevention of cardiovascular diseases is a top priority in countries with limited health system budgets such as Iran.

Eighty seven to hundred percent of patients dying from CVDs have at least one risk factor for cardiovascular diseases. Therefore, risk factor modification might prevent death and is a main priority. Combination drug therapy has been proposed as a cost-effective measure to reduce modifiable risk factors for cardiovascular disease. It has been showed that combination drug therapy can potentially decrease ischemic heart events and strokes by 88 and 80 percent, respectively.

The study is designed as a pragmatic cluster randomized controlled trial. The purpose of this study is to determine the effects of a fixed dose combination of either enalapril or valsartan, with hydrochlorthiazide, atorvastatin and acetylsalicylic acid (PolyPill) on primary and secondary prevention of cardiovascular disease in Iranian adults older than 50. Two formulations of Polypill tablets were used. The first formulation (Polypill-E) contained enalapril 5 mg. If participants developed cough, they were switched by a trained physician to Polypill-V, containing valsartan 40 mg instead of enalapril.

The investigators have previously tested the same combination in a different setting in Golestan, Northeast of Iran. The results of the study were published in the Lancet. The current study enrolls participants of Pars Cohort running in Fars province, southern Iran, aged above 50. A total of 4415 participants (91 clusters) were recruited following inclusion and exclusion criteria. The study comprises two arms as follows:

2200 randomly selected participants receive PolyPill tablets once daily and minimal care (which consists of direct education and pamphlet on cardiovascular risk reduction).

2215 randomly selected participants receive only minimal care as described above.

Endpoints include major cardiovascular events (MCVE).

ELIGIBILITY:
Inclusion Criteria:

* 50-79 years old
* Enrollment in the Pars Cohort Study

Exclusion Criteria:

1. Not consenting to participate in the study
2. Hypersensitivity to any of PolyPill components:

   1. Hypersensitivity to Non-steroidal anti-inflammatory agents
   2. Hypersensitivity to statins
   3. Hypersensitivity to hydrochlorothiazide or sulfonamides
   4. Hypersensitivity to enalapril and valsartan
3. Past medical history of angioedema
4. Medical history of GI bleeding or peptic ulcer in the last 3 months
5. Pregnancy or lactation
6. Bleeding disorders such as hemophilia
7. Receiving regular anticoagulation therapy
8. Alcohol consumption greater than 40gr/week
9. Advanced liver disease
10. Uncontrolled seizures
11. Asthma with any of the following criteria present:

    1. Daily symptoms
    2. Asthmatic attacks waking the patient from sleep more than once a week
    3. History of nasal polyps
    4. Aspirin sensitive asthma
    5. Presence of rhinitis symptoms not due to infection
12. Past medical history of gout
13. Serum creatinine values above 2 mg/dL
14. Glomerular Filtration Rate (GFR) below 30 mL/min
15. Hemoglobin concentrations below 11 g/dL for males and 10 g/dL for females
16. BP < 90/60 mmHg
17. Debilitating medical/mental disorders affecting compliance (including psychosis, disabilities, and blindness)
18. Past medical history of stroke

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4415 (Actual)
Dates: Start 2015-12-20 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
Major Cardiovascular Events (MCVE) | 5 years
  the first occurrence of acute coronary syndrome (non-fatal myocardial infarction and unstable angina), fatal myocardial infarction, sudden cardiac death, new-onset heart failure, coronary artery revascularization procedures, transient ischemic attack, cerebrovascular accidents (fatal or non-fatal), and hospitalization due to any of the mentioned conditions.

SECONDARY OUTCOMES:
Number of Subjects Developing Adverse Events | 5 years
  Number of participants who experience adverse effects to the PolyPill tablet leading to discontinuation
Compliance | 5 years
  Compliance is measured by pill-count in participants of the intervention arm as percent pills taken
Non cardiovascular mortality | 5 years
  Any death other than those due to CVDs during 5 years
Level of fasting blood sugar (mg/dL) | 5 years
  Changes in fasting blood sugar after 5 years
Level of blood pressure (mmHg) | 5 years
  Changes in blood pressure after 5 years
Level of total cholesterol (mg/dL) | 5 years
  Changes in total cholesterol after 5 years
Level of HDL (mg/dL) | 5 years
  Changes in HDL after 5 years
Level of LDL (mg/dL) | 5 years
  Changes in LDL after 5 years
Level of triglycerides (mg/dL) | 5 years
  Changes in triglycerides after 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, MD, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Pars Cohort Center, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roshandel G, Khoshnia M, Poustchi H, Hemming K, Kamangar F, Gharavi A, Ostovaneh MR, Nateghi A, Majed M, Navabakhsh B, Merat S, Pourshams A, Nalini M, Malekzadeh F, Sadeghi M, Mohammadifard N, Sarrafzadegan N, Naemi-Tabiei M, Fazel A, Brennan P, Etemadi A, Boffetta P, Thomas N, Marshall T, Cheng KK, Malekzadeh R. Effectiveness of polypill for primary and secondary prevention of cardiovascular diseases (PolyIran): a pragmatic, cluster-randomised trial. Lancet. 2019 Aug 24;394(10199):672-683. doi: 10.1016/S0140-6736(19)31791-X. PMID 31448738
- [Background] Malekzadeh F, Marshall T, Pourshams A, Gharravi M, Aslani A, Nateghi A, Rastegarpanah M, Khoshnia M, Semnani S, Salahi R, Thomas GN, Larijani B, Cheng KK, Malekzadeh R. A pilot double-blind randomised placebo-controlled trial of the effects of fixed-dose combination therapy ('polypill') on cardiovascular risk factors. Int J Clin Pract. 2010 Aug;64(9):1220-7. doi: 10.1111/j.1742-1241.2010.02412.x. PMID 20653798
- [Background] Ostovaneh MR, Poustchi H, Hemming K, Marjani H, Pourshams A, Nateghi A, Majed M, Navabakhsh B, Khoshnia M, Jaafari E, Mohammadifard N, Malekzadeh F, Merat S, Sadeghi M, Naemi M, Etemadi A, Thomas GN, Sarrafzadegan N, Cheng KK, Marshall T, Malekzadeh R. Polypill for the prevention of cardiovascular disease (PolyIran): study design and rationale for a pragmatic cluster randomized controlled trial. Eur J Prev Cardiol. 2015 Dec;22(12):1609-17. doi: 10.1177/2047487314550803. Epub 2014 Sep 17. PMID 25230980
- [Background] Lonn E, Bosch J, Teo KK, Pais P, Xavier D, Yusuf S. The polypill in the prevention of cardiovascular diseases: key concepts, current status, challenges, and future directions. Circulation. 2010 Nov 16;122(20):2078-88. doi: 10.1161/CIRCULATIONAHA.109.873232. No abstract available. PMID 21098469
- [Background] Malekzadeh F, Pourshams A, Marshall T. The preventive polypill--much promise, insufficient evidence. Arch Iran Med. 2007 Jul;10(3):430-1. No abstract available. PMID 17604490
- [Background] Majed M, Moradmand Badie S. A pilot double-blind randomised placebo-controlled trial of the effects of fixed-dose combination therapy ('polypill') on cardiovascular risk factors. Arch Iran Med. 2011 Jan;14(1):78-80. No abstract available. PMID 21194270
- [Background] PILL Collaborative Group; Rodgers A, Patel A, Berwanger O, Bots M, Grimm R, Grobbee DE, Jackson R, Neal B, Neaton J, Poulter N, Rafter N, Raju PK, Reddy S, Thom S, Vander Hoorn S, Webster R. An international randomised placebo-controlled trial of a four-component combination pill ("polypill") in people with raised cardiovascular risk. PLoS One. 2011;6(5):e19857. doi: 10.1371/journal.pone.0019857. Epub 2011 May 25. PMID 21647425
- [Background] Yusuf S, Pais P, Sigamani A, Xavier D, Afzal R, Gao P, Teo KK. Comparison of risk factor reduction and tolerability of a full-dose polypill (with potassium) versus low-dose polypill (polycap) in individuals at high risk of cardiovascular diseases: the Second Indian Polycap Study (TIPS-2) investigators. Circ Cardiovasc Qual Outcomes. 2012 Jul 1;5(4):463-71. doi: 10.1161/CIRCOUTCOMES.111.963637. Epub 2012 Jul 10. PMID 22787067
- [Background] Indian Polycap Study (TIPS); Yusuf S, Pais P, Afzal R, Xavier D, Teo K, Eikelboom J, Sigamani A, Mohan V, Gupta R, Thomas N. Effects of a polypill (Polycap) on risk factors in middle-aged individuals without cardiovascular disease (TIPS): a phase II, double-blind, randomised trial. Lancet. 2009 Apr 18;373(9672):1341-51. doi: 10.1016/S0140-6736(09)60611-5. Epub 2009 Mar 30. PMID 19339045
- [Background] Wald NJ, Law MR. A strategy to reduce cardiovascular disease by more than 80%. BMJ. 2003 Jun 28;326(7404):1419. doi: 10.1136/bmj.326.7404.1419. PMID 12829553
- [Derived] Malekzadeh F, Gandomkar A, Poustchi H, Etemadi A, Roshandel G, Attar A, Abtahi F, Sadeghi Boogar S, Mohammadkarimi V, Fattahi MR, Mohagheghi A, Malekzadeh R, Sepanlou SG. Effectiveness of polypill for primary and secondary prevention of cardiovascular disease: a pragmatic cluster-randomised controlled trial (PolyPars). Heart. 2024 Jun 25;110(14):940-946. doi: 10.1136/heartjnl-2023-323614. PMID 38485210
- [Derived] Malekzadeh F, Gandomkar A, Malekzadeh Z, Poustchi H, Moghadami M, Fattahi MR, Moini M, Anushiravani A, Mortazavi R, Sadeghi Boogar S, Mohammadkarimi V, Abtahi F, Merat S, Sepanlou SG, Malekzadeh R. Effectiveness of Polypill for Prevention of Cardiovascular Disease (PolyPars): Protocol of a Randomized Controlled Trial. Arch Iran Med. 2020 Aug 1;23(8):548-556. doi: 10.34172/aim.2020.58. PMID 32894967